CLINICAL TRIAL: NCT05788562
Title: The Relevance Between the Level of Fetal Hemoglobin and Short-term Complications in Extremely Preterm Infants
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: wu hui
Record Dates: First submitted 2023-03-15; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2022-06

CONDITIONS: Fetal Hemoglobin
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: Incorporate blood gas analysis indicators in D1-D7, after birth,1 week before and on the day of onset of early complications
- Control group: Incorporate blood gas analysis indicators in D1-D7,D14,D28after birth and the day of diacharge

SUMMARY:
A monocentric prospective study was conducted to find the relevance between the level of fetal hemoglobin and short-term complications in extremely preterm infants

ELIGIBILITY:
Inclusion Criteria:

1. Preterm infants with gestational age <32 weeks or birth weight <1500g
2. Parents agree to attend

Exclusion Criteria:

1. serious functional or organic diseases
2. severe congenital deformity
3. parents reject to attend

Ages: 1 Day to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants with gestational age <32 weeks or birth weight <1500g
Sampling Method: Non-Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-02-18 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence and severity of early complications in premature infants | 2022.1-2023.1
  include necrotizing enterocolitis,bronchopulmonary dysplasia,retinopathy, Intraventricular hemorrhage above degree Ⅱ,leukomalacia,late-onset sepsis

CONTACTS AND LOCATIONS:
Locations (1):
- First hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No